CLINICAL TRIAL: NCT07310030
Title: Immediate Effects of Neuro-Athletic Training on Physical Fitness Parameters in Young Individuals
Brief Title: Neuro-Athletic Training Effects in Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Beyza Tanrıöğen, research assistant, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Istinye BT 3
Record Dates: First submitted 2025-11-22; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Health Young Individuals; Physical Fitness
Keywords: neuro-athletic training; saccadic eye movements; sports related performance; physical fitness
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuro-athletic training programme (Stretching, Balance Training, Vertical Jump and Eye Exercise) (Experimental): Neuro-athletic training programme (Stretching, Balance Training, Vertical Jump and Eye Exercise)
  This group group will perform all exercises included in the control group, with the addition of eye exercises. In addition to the control group protocol, participants in this group will complete various video-based eye exercises, including smooth pursuit, saccadic movements, and anti-saccade tasks. Furthermore, the Brock string exercise will be administered to train depth perception.
  All exercises in the program are implemented as part of a warm-up routine to help prevent injuries and pose no health risks for healthy individuals. If symptoms such as dizziness or visual fatigue occur during the eye exercises, the session will be terminated. All exercises will be performed under the supervision of a physiotherapist to ensure correct execution and safety. The warm-up duration will be kept equal for both groups.
  Interventions: Behavioral: Experimental: Neuro-athletic training programme (Stretching, Balance Training, Vertical Jump and Eye Exercise)
- Stretching, Balance Training and Vertical Jump Exercise Program (without eye exercises) (Active Comparator): Stretching, Balance Training and Vertical Jump Exercise Program (without eye exercises)
  This group (control) group will perform only stretching exercises, balance training, and vertical jump exercises. Stretching exercises will consist of static stretches targeting the hip flexors, hamstrings, quadriceps, and gastrocnemius muscle groups, with each position held for 20-30 seconds for two repetitions. Balance training will be performed on a Both Sides Utilized ball and balance board in a single-leg stance, with three trials for each leg; each trial will last 15 seconds, with 30 seconds of rest between trials.
  All exercises are incorporated into a warm-up program to help prevent injuries and pose no health risks for healthy individuals. All exercises will be performed under the supervision of a physiotherapist to ensure correct execution and control. No eye exercises will be administered to the control group. The warm-up duration will be kept equal for both groups.
  Interventions: Behavioral: Active Comparator: Stretching, Balance Training and Vertical Jump Exercise Program (without eye exercises) Control group

INTERVENTIONS:
Behavioral: Experimental: Neuro-athletic training programme (Stretching, Balance Training, Vertical Jump and Eye Exercise) — Neuro-athletic training programme (Stretching, Balance Training, Vertical Jump and Eye Exercise)
  This group group will perform all exercises included in the control group, with the addition of eye exercises. In addition to the control group protocol, participants in this group will complete various video-based eye exercises, including smooth pursuit, saccadic movements, and anti-saccade tasks. Furthermore, the Brock string exercise will be administered to train depth perception.
  All exercises in the program are implemented as part of a warm-up routine to help prevent injuries and pose no health risks for healthy individuals. If symptoms such as dizziness or visual fatigue occur during the eye exercises, the session will be terminated. All exercises will be performed under the supervision of a physiotherapist to ensure correct execution and safety. The warm-up duration will be kept equal for both groups.
  Arms: Neuro-athletic training programme (Stretching, Balance Training, Vertical Jump and Eye Exercise)
Behavioral: Active Comparator: Stretching, Balance Training and Vertical Jump Exercise Program (without eye exercises) Control group — Stretching, Balance Training and Vertical Jump Exercise Program (without eye exercises)
  This group (control) group will perform only stretching exercises, balance training, and vertical jump exercises. Stretching exercises will consist of static stretches targeting the hip flexors, hamstrings, quadriceps, and gastrocnemius muscle groups, with each position held for 20-30 seconds for two repetitions. Balance training will be performed on a Both Sides Utilized ball and balance board in a single-leg stance, with three trials for each leg; each trial will last 15 seconds, with 30 seconds of rest between trials.
  All exercises are incorporated into a warm-up program to help prevent injuries and pose no health risks for healthy individuals. All exercises will be performed under the supervision of a physiotherapist to ensure correct execution and control. No eye exercises will be administered to the control group. The warm-up duration will be kept equal for both groups.
  Arms: Stretching, Balance Training and Vertical Jump Exercise Program (without eye exercises)

SUMMARY:
This study aims to examine the acute effects of a single session of neuro-athletic training (NAT) on key physical fitness parameters in young adults. Neuro-athletic training is a contemporary approach that integrates neuroscience principles with athletic conditioning, focusing not only on muscular strength but also on optimizing the interaction between the nervous system and the musculoskeletal system. By targeting visual, vestibular, and proprioceptive mechanisms, NAT seeks to enhance motor output, coordination, movement efficiency, and decision-making processes.

Although NAT has gained increasing attention in sports performance programs, most existing research has focused on long-term training adaptations in elite athletes. Evidence regarding its immediate effects-especially in healthy university-aged individuals-is still limited. Preliminary findings suggest that exercises incorporating cognitive load and sensory integration may improve various aspects of performance; however, the short-term influence of NAT on balance, flexibility, reaction time, and power has not been fully clarified.

In this context, the present controlled experimental study compares the effects of a single NAT session with those of a traditional warm-up routine. The study evaluates acute changes in balance, flexibility, vertical power, and reaction time to determine whether NAT can produce immediate performance benefits. The findings are expected to contribute to a clearer understanding of how neuro-athletic principles can be integrated into preparatory exercise routines to enhance both neuromuscular and cognitive-motor performance in young adults.

DETAILED DESCRIPTION:
Our study is designed as a randomized, controlled, single-blind trial. Participants will be randomly assigned to two groups (intervention group, n=11; control group, n=11) following a pre-test-intervention-post-test design.

Control Group Exercises

The control group will perform only stretching exercises, balance training, and vertical jump exercises. Stretching exercises will include static stretches targeting the hip flexors, hamstrings, quadriceps, and gastrocnemius muscle groups, with each position held for 20-30 seconds for two repetitions. Balance training will be performed on a Both Sides Utilized ball and balance board in a single-leg stance, with three trials for each leg; each trial will last 15 seconds with 30 seconds of rest between trials. These exercises are incorporated into a warm-up routine to help prevent injuries and pose no health risks for healthy individuals. All exercises will be conducted under the supervision of a physiotherapist to ensure proper execution and safety. No eye exercises will be administered to the control group. The duration of the warm-up will be kept equal for both groups.

Intervention Group Exercises

The intervention group will perform all exercises included in the control group, in addition to eye exercises. Along with the control group protocol, the intervention group will complete video-based eye exercises, including smooth pursuit, saccadic eye movements, and anti-saccade tasks. Additionally, the Brock string exercise will be used to train depth perception. These exercises are included as part of the warm-up program to help prevent injuries and are considered safe for healthy individuals. If symptoms such as dizziness or visual fatigue occur during the eye exercises, the session will be terminated. All exercises will be conducted under the supervision of a physiotherapist to ensure correct performance and safety. The warm-up duration will be kept equal for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults aged 18-35 years
* Not participating in professional sports
* No visual impairments
* Provide written informed consent and agree to participate in the study

Exclusion Criteria:

* Diagnosed musculoskeletal disorder
* Diagnosed neurological or orthopedic condition
* Balance disorders (e.g., vestibular system problems, frequent dizziness)
* History of serious musculoskeletal injury or surgery within the past 6 months
* Unable to perform the exercises during assessment due to pain

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Flexibility Test: Sit and Reach | 4 weeks
  The Sit and Reach test will be applied solely to assess participants' flexibility. Participants will sit on a flat surface with legs extended, arms and fingers stretched forward. They will bend the torso forward and hold the farthest reachable point for 1-2 seconds. Three trials will be performed, and the best score will be recorded. This test is a valid and reliable method for flexibility assessment.
Balance Assessment | 4 weeks
  Dynamic and static balance will be objectively assessed in a standing position using the TecnoBody® system. The system will measure the center of pressure, path length, and the sway area of the center of pressure. Lower sway values indicate better lower extremity stability and balance ability.

SECONDARY OUTCOMES:
Fukuda Stepping Test | 4 weeks
  The Fukuda Stepping Test will be used to evaluate the integrity of the vestibulospinal reflex. Participants will be asked to march in place for 50 steps with eyes closed and arms extended forward at shoulder height on a firm surface. The deviation angle and displacement distance relative to the starting position will be recorded. A deviation greater than 30 degrees may indicate asymmetry in the vestibular system.
Upper Extremity Reaction Time | 4 weeks
  Upper extremity reaction time will be measured similarly, using the hands to touch the lights. Each measurement will be repeated three times, with the best score used for analysis. The device has been shown to be valid and reliable for measuring both lower and upper extremity reaction times.
Lower Extremity Reaction Time | 4 weeks
  Lower extremity reaction time will be assessed using the BlazePod™ device. Participants will balance on one leg and attempt to touch randomly illuminated lights with their foot for 30 seconds.
Vertical Jump Test | 4 weeks
  Participants will first stand on a flat surface to determine their maximum reach with extended arms, then perform a vertical jump from a squat position, reaching the highest point with their fingertips. Three trials will be conducted, and the highest value will be recorded. Jump height reflects lower extremity power output.
Saccadic Eye Movement Assessment | 4 weeks
  Participants will sit on a stable chair with their head kept as still as possible. The assessor will hold one pen or visual target in each hand, positioned at eye level with 15-20° spacing. Participants will move their eyes rapidly and accurately between the targets, without moving their head. The test will be performed in both horizontal and vertical planes. This is a valid method to assess visual-motor control and saccadic eye movement speed.
Demographic Data | 4 weeks
  Participants' demographic data will be collected such as age
weigh | 4 weeks
  Participants' demographic data will be collected such as weight
height | 4 weeks
  Participants' demographic data will be collected such as height.

IPD SHARING:
Plan to Share IPD: No